CLINICAL TRIAL: NCT00285779
Title: A Double-Blind, Randomized, Multicenter Pilot Study to Evaluate the Efficacy and Safety of Etanercept 50mg SC Twice Weekly in the Treatment of Moderate to Severe Lichen Planus
Brief Title: Use of Etanercept in the Treatment of Moderate to Severe Lichen Planus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Stanford University (Other)
Collaborators: Wright State University (Other); Tufts Medical Center (Other); University of Louisville (Other); Wake Forest University Health Sciences (Other); University of Michigan (Other); Emory University (Other); University Hospitals Cleveland Medical Center (Other); Icahn School of Medicine at Mount Sinai (Other); Oregon Health and Science University (Other); The Cleveland Clinic (Other); Fivenson, David, M.D. (Individual)
Responsible Party: Principal Investigator, David Fiorentino, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20041132; NCT00568581 (obsolete NCT alias); NCT00691106 (obsolete NCT alias)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Lichen Planus
MeSH Terms: conditions — Lichen Planus | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo injection (Placebo Comparator): patients receive normal saline injection twice weekly for weeks 1-12
  Interventions: Drug: Placebo
- Etanercept (Experimental): patients receive etanercept injection twice weekly for weeks 1-12.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — etanercept 50 mg twice weekly for 12 weeks
  Other Names: Enbrel
  Arms: Etanercept
Drug: Placebo
  Arms: Placebo injection

SUMMARY:
The purpose is to assess the response of subjects to etanercept (as compared to placebo) in treating the physical signs of mucosal and cutaneous lichen planus. The investigators also wish to assess the effect of etanercept on disease-related itching, pain, and serious adverse events in patients with lichen planus.

DETAILED DESCRIPTION:
Lichen planus affects up to 1% of the worldwide population. Recent estimates suggest approximately 0.44% of the US population suffers from this disease. Oral or genital involvement occurs in 60-70% of patients, and it may be the sole manifestation of disease in 20-30% of patients.

Lichen planus is a mucocutaneous disorder that can involve the skin, oral or genital mucosa, conjunctiva, and nails. On the skin, the disease presents as multiple papules, which can be localized or generalized, that are often extremely itchy. Mucosal disease can consist of either asymptomatic plaques or extremely painful erosive lesions. The disease course is unpredictable and typically lasts 1-2 years but can follow a chronic, relapsing course. Erosive mucosal disease is important to aggressively treat for many reasons: First, the associated pain can be debilitating for the patient. Patients with severe oral lichen planus can become malnourished due to pain associated with eating. Vulvar disease can cause dyspareunia, burning pain, and discharge; second, the disease tends to be chronic, with little chance for self-resolution; third, erosive disease is associated with an increased risk of squamous cell carcinoma in the affected areas. These cancers occur in up to 1% of patients over a 3-year period, and they can be aggressive and even-life threatening for the patient if not recognized and treated early.

Several lines of evidence suggest that TNF-alpha plays a role in the pathogenesis of lichen planus. It has been shown that there are increased levels of TNF-alpha in the serum of these patients. In addition, skin and mucosal biopsies show increased TNF-alpha produced by the infiltrating lymphocytes as well as the basal keratinocytes. It has been suggested that the expression of TNF-alpha receptor on the basal keratinocytes may contribute to apoptosis. Also, TNFR1 (a TNF-alpha receptor) is expressed by the infiltrating mononuclear cells as well as the keratinocytes. Increased levels of soluble TNF receptors are also found in the serum of patients with lichen planus. A recent report also has shown that polymorphisms in the TNF-alpha gene are associated with both oral and cutaneous lichen planus. Finally, thalidomide, which partly functions as a potent inhibitor of TNF-alpha transcription, has been shown to be effective (in small case series and reports) in selected patients for the treatment of oral and genital lichen planus. However, thalidomide is a potent teratogen and cannot be used in women of childbearing potential. In addition, thalidomide usage not uncommonly results in neurotoxicity, which can be permanent, and thus limits use of this drug. Despite the evidence for a role of TNF-alpha in LP there are no reports of any TNF inhibitors being used for this disease.

This is a double-blind, placebo-controlled pilot study to observe the safety and efficacy of etanercept in patients with lichen planus.

This study will consist of 3 periods: first, a double-blind period (weeks 0-12) in which subjects will be randomized to etanercept 50 mg twice weekly or placebo; second, an open-label period (weeks 12-24) in which subjects who were randomized to placebo treatment, who have not achieved a complete remission, will be rolled over to use etanercept at 50 mg twice weekly. Subjects who previously received etanercept during weeks 0-12, who have not achieved a complete remission, will be continued on etanercept at a lower dosage of 25 mg twice weekly for weeks 12-24; third, an 8 week follow-up period for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Must carry a diagnosis of lichen planus as determined by biopsy
* Patients must have a score of 3 or greater on the physician global assessment (PGA).
* Patient must be considered appropriate for systemic therapy based upon fulfilling one of the following criteria:

  1. inability to maintain weight due to pain with eating, chewing, or swallowing;
  2. dyspareunia or dysuria due to genital lesions;
  3. itch/pain of sufficient severity that activities of daily living are significantly affected
* Must be off systemic lichen planus treatment for 4 weeks prior to starting etanercept
* If using topical corticosteroid to the affected areas, the dose and frequency must be unchanged for 2 weeks prior to beginning the study agent and during the course of the study.
* Must be off topical cyclosporine, tacrolimus, or pimecrolimus for 2 weeks prior to starting the study drug and for the entire duration of the study.
* Must be able and willing to give written informed consent and comply with the requirements of the study protocol and must authorize release and use of protected health information.
* Women of childbearing potential must have a negative pregnancy test at the time of entry into the study and must be practicing successful contraception for at least 3 months prior to the study.
* Subject or designee must have the ability to self-inject investigational product.
* Screening laboratory results are within the following parameters:

  * Hemoglobin > 10 g/dL
  * White blood cells > 3.5 x 10^9/L
  * Neutrophils > 1.5 x 10^9/L
  * Platelets > 100 x 10^9/L
  * Lymphocytes > 0.5 x 10^9/L
  * Serum creatinine < 1.5 mg/dL
  * Hepatitis C serology - nonreactive
  * AST and ALT < 2X upper limit of normal (ULN)

Exclusion Criteria:

* Subject is currently enrolled in another investigational device or drug trial(s), or subject has received investigational agent(s) within 90 days of baseline visit.
* Known HIV-positive status, any other immuno-suppressive disease, or inability to practice safe sex during the length of the study
* Subject has been diagnosed with a malignancy within the past 5 years
* Subject has signs or symptoms of a lymphoproliferative disease.
* Other skin or mucosal disease that might interfere with lichen planus assessments.
* Lichen planus variants including hypertrophic, atrophic, follicular (including lichen planopilaris), and bullous cutaneous forms.
* Patients with lichen sclerosis et atrophicus (LS&A)
* Clinical history and lesion distribution suspicious for a lichenoid drug eruption
* Severe co-morbidities
* History of tuberculosis (TB) or positive PPD at screening. Known history of active hepatitis B or C, or lupus, SLE, history of multiple sclerosis or prior episode of central nervous system demyelination, transverse myelitis, optic neuritis, epilepsy, psychiatric condition, or other chronic serious medical illnesses.
* Subject has a diagnosis of congestive heart failure (CHF) of any severity
* Use of a live vaccine 90 days prior to, or during this study.
* Previous exposure and/or known sensitivity to etanercept
* Concurrent use, or failure of, any TNF-inhibitor
* Previous exposure to alefacept or efalizumab within 6 weeks of administration of study drug
* Concurrent sulfasalazine therapy
* Prior or concurrent cyclophosphamide therapy
* Active severe infections, or prior infection requiring hospitalization or oral/intravenous antibiotics within 4 weeks before screening visit, or between the screening and baseline visits.
* Active inflammatory bowel disease or peptic ulcer disease
* Drug or alcohol abuse within 12 months of screening visit.
* History of non-compliance with other therapies
* Pregnant or lactating
* Documented presence of any of the following:

  * Proteinuria > 1+ by dipstick screening
  * 24 Hour protein excretion > 0.5 g
  * Symptomatic liver disease with serum albumin < 3 G/DL
  * PT or PTT > ULN, or
  * Chronic liver disease
* Documented forced vital capacity < 50% of predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Fiorentino, MD, PhD, Principal Investigator — Stanford University; David F Fiorentino, MD, PhD, Study Director — Stanford University
Locations (12):
- United States (12):
  - Stanford University Medical Center, Stanford, California
  - Emory University, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Tufts - New England Medical Center, Boston, Massachusetts
  - David Fivenson, M.D. Dermatology, PLLC, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Wright State University School of Medicine, Dayton, Ohio
  - Oregon Health & Science University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, multi-center interventional trial in which patients were recruited at 11 sites in the United States (10 academic and one private practice). Enrollment was between June, 2006 and December, 2008. The first subject was enrolled in August, 2006 and the last patient was enrolled in November, 2008.
Groups:
- Placebo Injection: Placebo: Normal saline twice weekly for 12 weeks
Period: Placebo-controlled Period (wk 1-12)
Arm/Group | Placebo Injection | Etanercept
Started | 14 | 13
Completed | 11 | 12
Not Completed | 3 | 1
Period: Open Label Period (wk 12-24)
Arm/Group | Placebo Injection | Etanercept
Started | 11 | 12
Completed | 9 | 10
Not Completed | 2 | 2
Period: Follow-up Period (wk 24-32)
Arm/Group | Placebo Injection | Etanercept
Started | 9 | 10
Completed | 8 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Injection | Etanercept | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (16.9) | 57.4 (16.0) | 53.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Achieving a Response in Mucosal Disease (or Cutaneous Disease if no Mucosal Disease) at 12 Weeks
Description: Physician global assessment of disease scores: 0=clear; 1=minimal disease; 2=mild disease; 3=moderate disease; 4=severe disease. Subjects had a level >=3 at baseline. To be considered a responder, the subject must achieve a level of 0 or 1, or, at least a 2 point improvement in the scale.
Time Frame: 12 weeks
Population: Intention to treat analysis (all participants received at least one dose of study drug). Missing data imputed using Last Observation Carried Forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
percentage of participants | 28.6 | 0
Statistical Analysis 1: Comparison: Placebo Injection vs Etanercept; Test type: Superiority or Other; p = 0.0978, Fisher Exact

2. Secondary Outcome: Count of Patients Achieving a Response in Cutaneous or Mucosal Disease at 24 Weeks
Description: as for outcome 1
Time Frame: Baseline; Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
Participants | 5 | 4
Statistical Analysis 1: Comparison: Placebo Injection vs Etanercept; Test type: Other; p > 0.9999, Fisher Exact

3. Secondary Outcome: The Physician Assessment of Surface Area of Disease (PSAD) for Oral Disease at 12 and 24 Weeks
Description: The percentage of surface area involved with disease is reported as assessed by the physician using a Likert scale. Assessment scores range from 0-5, with lower scores corresponding lower percentage of surface area with disease. 0=clear, 1=<2%, 2=2-9%, 3=10-29%, 4=30-50%, 5=>50%.
Time Frame: Baseline; Week 12; Week 24
Population: Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 13 | 13
  Baseline | 1.2 (1.31) | 1.6 (1.73)
  Week 12: number analyzed (Participants) | 11 | 12
  Week 12 | 0.8 (1.03) | 1.5 (1.44)
  Week 24: number analyzed (Participants) | 9 | 10
  Week 24 | 1.1 (1.10) | 1.5 (1.20)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.031, Wilcoxon Paired
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.34, Wilcoxon Paired
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.13, Wilcoxon Paired
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.22, Wilcoxon Paired

4. Secondary Outcome: The Physician Assessment of Surface Area of Disease (PSAD) for Genital Disease at 12 and 24 Weeks
Description: as for outcome 3
Time Frame: Baseline; Week 12; Week 24
Population: Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 13 | 13
  Baseline | 0.3 (0.82) | 0.4 (1.33)
  Week 12: number analyzed (Participants) | 12 | 12
  Week 12 | 0.5 (0.96) | 0.4 (1.38)
  Week 24: number analyzed (Participants) | 9 | 10
  Week 24 | 0.7 (1.05) | 0.5 (1.50)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p > 0.9999, Wilcoxon Paired
Statistical Analysis 2: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p > 0.9999, Wilcoxon Paired

5. Secondary Outcome: The Physician Assessment of Surface Area of Disease (PSAD) for Skin Disease at 12 and 24 Weeks
Description: as for outcome 3
Time Frame: Baseline; Week 12; Week 24
Population: Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 13 | 13
  Baseline | 2.8 (1.56) | 1.8 (1.61)
  Week 12: number analyzed (Participants) | 12 | 12
  Week 12 | 2.2 (1.77) | 1.7 (1.43)
  Week 24: number analyzed (Participants) | 9 | 10
  Week 24 | 1.0 (0.94) | 1.6 (1.36)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.25, Wilcoxon Paired
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p > 0.9999, Wilcoxon Paired
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.063, Wilcoxon Paired
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p > 0.9999, Wilcoxon Paired

6. Secondary Outcome: Cutaneous Target Lesion Scores - Erythema, at 12 and 24 Weeks
Description: This is an investigator-based assessment of a single preselected target skin lesion. Assessment scores range from 0-3 on a Likert scale, with higher scores meaning worse erythema. 0=clear, 1=mild/pink, 2=moderately red, 3=severely red/violaceous.
Time Frame: Week 12; Week 24
Population: Participants with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 12 | 9
  Baseline | 2.5 (0.76) | 2.3 (0.67)
  Week 12: number analyzed (Participants) | 11 | 8
  Week 12 | 1.6 (1.30) | 1.8 (0.83)
  Week 24: number analyzed (Participants) | 8 | 8
  Week 24 | 0.9 (1.05) | 1.8 (0.97)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.063, Wilcoxon Paired
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.25, Wilcoxon Paired
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.031, Wilcoxon Paired
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.32, Wilcoxon Paired

7. Secondary Outcome: Cutaneous Target Lesion Scores - Elevation, at 12 and 24 Weeks
Description: This is an investigator-based assessment of a single preselected target skin lesion. Assessment scores range from 0-3 on a Likert scale, with higher scores meaning worse elevation. 0=flat, 1=barely palpable (<0.5 mm), 2=moderate (0.5 mm-1 mm), 3=severe (>1 mm).
Time Frame: Week 12; Week 24
Population: Participants with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 12 | 9
  Baseline | 2.1 (0.64) | 2.1 (0.87)
  Week 12: number analyzed (Participants) | 11 | 8
  Week 12 | 1.5 (1.16) | 1.6 (0.70)
  Week 24: number analyzed (Participants) | 8 | 8
  Week 24 | 1.0 (1.22) | 0.8 (0.83)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.094, Wilcoxon Paired
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.25, Wilcoxon Paired
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.13, Wilcoxon Paired
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.13, Wilcoxon Paired

8. Secondary Outcome: Cutaneous Target Lesion Scores - Scale, at 12 and 24 Weeks
Description: This is an investigator-based assessment of a single preselected target skin lesion. Assessment scores range from 0-3 on a Likert scale, with higher scores meaning worse scaling. 0=none, 1=fine/dusty scale, 2=moderate scale, 3=thick/tenacious scale.
Time Frame: Week 12; Week 24
Population: Participants with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 12 | 9
  Baseline | 0.9 (0.76) | 1.2 (0.79)
  Week 12: number analyzed (Participants) | 11 | 8
  Week 12 | 0.8 (0.72) | 0.8 (0.66)
  Week 24: number analyzed (Participants) | 8 | 8
  Week 24 | 0.4 (0.99) | 0.8 (0.83)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.63, Wilcoxon Paired
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.38, Wilcoxon Paired
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.38, Wilcoxon Paired
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.50, Wilcoxon Paired

9. Secondary Outcome: Cutaneous Target Lesion Scores - Total, at 12 and 24 Weeks
Description: This score sums all of the 3 elements of the target lesion score (erythema, elevation, scale) described in Outcome Measures 6-8. Assessment scores range from 0-9 on a Likert scale, with higher numbers meaning more severe disease in the target skin lesion.
Time Frame: Week 12; Week 24
Population: Participants with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 12 | 9
  Baseline | 4.7 (2.55) | 3.9 (3.02)
  Week 12: number analyzed (Participants) | 11 | 8
  Week 12 | 3.1 (3.10) | 2.5 (2.50)
  Week 24: number analyzed (Participants) | 8 | 8
  Week 24 | 1.3 (2.52) | 2.4 (2.59)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.031, Wilcoxon Paired
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.094, Wilcoxon Paired
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.039, Wilcoxon Paired
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.19, Wilcoxon Paired

10. Secondary Outcome: Patient Assessment of Pain on a Visual Analogue Scale (VAS) at 12 and 24 Weeks
Description: Participants were asked to indicate their pain level by marking it on a 10 cm linear VAS scale. The number of centimeters from the left end of the line to the mark was measured in cm. Total range was 0-10. Lower scores correspond to less pain, higher scores correspond to more pain.
Time Frame: Baseline; Week 12; Week 24
Population: Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 13 | 13
  Baseline | 3.8 (3.08) | 3.4 (2.50)
  Week 12: number analyzed (Participants) | 12 | 13
  Week 12 | 3.4 (3.08) | 3.0 (2.85)
  Week 24: number analyzed (Participants) | 9 | 11
  Week 24 | 2.4 (2.83) | 2.8 (3.25)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.26, Paired t test
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.55, Paired t test
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.18, Paired t test
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.13, Paired t test

11. Secondary Outcome: Patient Assessment of Pruritus (Itching) on a Visual Analogue Scale (VAS) at 12 and 24 Weeks
Description: Participants were asked to indicate their itching level by marking it on a 10 cm linear VAS scale. The number of centimeters from the left end of the line to the mark was measured in cm. Total range was 0-10. Lower scores correspond to less itching, higher scores correspond to more itching.
Time Frame: Baseline; Week 12; Week 24
Population: Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 13 | 13
  Baseline | 3.8 (2.84) | 3.2 (2.55)
  Week 12: number analyzed (Participants) | 12 | 13
  Week 12 | 3.3 (3.38) | 3.4 (3.14)
  Week 24: number analyzed (Participants) | 9 | 11
  Week 24 | 1.5 (1.64) | 3.0 (2.71)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.51, Paired t test
Statistical Analysis 2: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.47, Paired t test
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.087, Paired t test
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.86, Paired t test

12. Secondary Outcome: Patient Assessment of Overall Disease Severity (Patient Global Assessment) at 12 and 24 Weeks
Description: Participants were asked to indicate their rate their overall assessment of disease severity compared to where it was at their baseline visit. The scale ranges from 0-5, with lower scores correspond to more disease improvement. 0=clear/no disease, 1=much improved (>75% improved), 2=improved (25-75%), 3=minimally improved (<25%), 4=no change, 5=worsened disease.
Time Frame: Baseline; Week 12; Week 24
Population: Participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline: number analyzed (Participants) | 9 | 10
  Baseline | 3.9 (0.87) | 4.1 (0.54)
  Week 12: number analyzed (Participants) | 8 | 10
  Week 12 | 2.3 (1.56) | 3.1 (1.23)
  Week 24: number analyzed (Participants) | 7 | 10
  Week 24 | 2.9 (1.46) | 2.6 (1.43)
Statistical Analysis 1: Comparison: Placebo Injection; Week 12 versus baseline; Test type: Other; p = 0.033, Paired t test
Statistical Analysis 2: Comparison: Etanercept; Week 12 versus baseline; Test type: Other; p = 0.069, Paired t test
Statistical Analysis 3: Comparison: Placebo Injection; Week 24 versus baseline; Test type: Other; p = 0.015, Paired t test
Statistical Analysis 4: Comparison: Etanercept; Week 24 versus baseline; Test type: Other; p = 0.026, Paired t test

13. Secondary Outcome: The Count of Subjects Experiencing Serious Adverse Events (SAEs) by Week 12 and Week 24
Description: A serious adverse event was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Baseline; Week 12; Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 14 | 13
Participants
  SAE by week 12 | 0 | 0
  SAE by week 24 | 0 | 1

14. Secondary Outcome: The Count of Placebo Patients Who do Not Have a Complete Response (Defined as a Physician Global Assessment of "Clear") at 12 Weeks
Description: A complete response is defined as a score of 0 (representing "no disease") on the Physician Global Assessment. Physician global assessment of disease scores: 0=clear; 1=minimal disease; 2=mild disease; 3=moderate disease; 4=severe disease. This endpoint is the number of patients on placebo that had any score other than 0 on this measure.
Time Frame: 12 weeks
Population: Only participants in the Placebo injection group were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Injection
Number analyzed (Participants) | 14
Participants | 13

15. Secondary Outcome: The Percentage of Placebo and Study-drug Patients Able to Discontinue Use of Topical Corticosteroids Through Week 24
Time Frame: 24 weeks
Population: Data were not collected for this outcome measure
Arm/Group | Placebo Injection | Etanercept
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This includes the entire 32 week timeframe of the trial. Thus, the placebo patients that cross over to etanercept from 12-24 weeks are also considered in the etanercept group during the 12-24 week timeframe. Also includes followup from 24-32 weeks.
Arm/Group | Placebo Injection | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/24
Other Adverse Events (participants affected / at risk) | 4/14 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=14) | Etanercept (N=24)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient hospitalized for 3 days with chest congestion and fever and later found to have pneumonia.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=14) | Etanercept (N=24)
Erythema at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Bruising at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Vaginal yeast infection (Infections and infestations) | 1 (1) | 2 (2)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Cataract surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Knee surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Gout flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
worsening diffuse joint pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Knee arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ankle and finger swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
increased back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Allergies (Immune system disorders) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
otitis media (Infections and infestations) | 0 (0) | 1 (1)
Oral pain with eating (Gastrointestinal disorders) | 1 (1) | 0 (0)
sore throat (Gastrointestinal disorders) | 0 (0) | 2 (2)
oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
facial flushing (Vascular disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
gastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
pruritis, generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial was terminated early due to low recruitment rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less